CLINICAL TRIAL: NCT00556868
Title: The Influence of Having Breakfast on Cognitive Performance and Mood in High School Students
Brief Title: The Influence of Having Breakfast on Cognitive Performance and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 241/2004
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Fasting
Keywords: High school students; Boarding school; Breakfast; Fasting; Memory; Attention; Mood
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Breakfast on the first day of intervention, fasting (no breakfast) on the second day of intervention
  Interventions: Other: Breakfast/no breakfast
- B (Experimental): Fasting (no breakfast) on the first day of intervention, breakfast on the second day of intervention
  Interventions: Other: Breakfast/no breakfast

INTERVENTIONS:
Other: Breakfast/no breakfast — A: Breakfast on the first day of intervention. Fasting (no breakfast) on the second day of intervention.
  B: Breakfast on the second day of intervention. Fasting (no breakfast) on the first day of intervention

SUMMARY:
Breakfast is often labelled the most important meal of the day.

Parents and teachers quite often stress its importance for successful learning during the morning hours. With declining numbers of children and especially adolescents eating breakfast regularly, the study examines the influence of breakfast consumption on cognition and mood of high school students.

ELIGIBILITY:
Inclusion Criteria:

* Healthy high school students

Exclusion Criteria:

* Diabetes

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2005-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Sustained attention, immediate memory, mood | 2 h

CONTACTS AND LOCATIONS:
Overall Officials: Katharina A Widenhorn-Mueller, PhD, Principal Investigator — Centre for Neuroscience and Learning, University of Ulm; Katrin Hille, PhD, Principal Investigator — Centre for Neuroscience and Learning, University of Ulm; Jochen Klenk, MPH, Principal Investigator — Institute of Epidemiology, University of Ulm; Weiland Ulrike, MD, Principal Investigator — Centre for Neuroscience and Learning, University of Ulm
Locations (1):
- Centre for Neuroscience and Learning, Ulm, Germany

REFERENCES:
- [Derived] Widenhorn-Muller K, Hille K, Klenk J, Weiland U. Influence of having breakfast on cognitive performance and mood in 13- to 20-year-old high school students: results of a crossover trial. Pediatrics. 2008 Aug;122(2):279-84. doi: 10.1542/peds.2007-0944. PMID 18676544